CLINICAL TRIAL: NCT04308343
Title: The Aromatase Inhibitor and Gnrh Antagonist Versus Methotrexate for Management of Undisturbed Ectopic Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali saber ali, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aromatase inhibitor in ectopic
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Methotrexate; Letrozole; cetrorelix

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Methotrexate group (Active Comparator)
  Interventions: Drug: Methotrexate
- Letrozole group (Active Comparator)
  Interventions: Drug: Letrozole
- Gonadotropins releasing hormone antagonist group (Active Comparator)
  Interventions: Drug: cetrotide

INTERVENTIONS:
Drug: Methotrexate — Drugs to treat undisturbed ectopic pregnancies
  Arms: Methotrexate group
Drug: Letrozole — Drugs to treat undisturbed ectopic pregnancies
  Arms: Letrozole group
Drug: cetrotide — Drugs to treat undisturbed ectopic pregnancies
  Arms: Gonadotropins releasing hormone antagonist group

SUMMARY:
The aim of this study is to :

1. Use of the aromatase inhibitor( letrozole) for the treatment of ectopic pregnancy compared to methotrexate.
2. Use of the Gnrh antagonist for the treatment of ectopic pregnancy compared to methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undisturbed ectopic pregnancy .Who are:

  1. have no significant pain
  2. have an unruptured tubal ectopic pregnancy with an adnexal mass smaller than 35mm with no visible heartbeat
  3. have a serum human chorionic gonadotropins level less than 1,500 IU/litre
  4. do not have an intrauterine pregnancy (as confirmed on an ultrasound scan) .

Exclusion Criteria:

1. An undisturbed ectopic pregnancy and significant pain
2. An undisturbed ectopic pregnancy with an adnexal mass of 35 mm or larger
3. An undisturbed ectopic pregnancy with a fetal heartbeat visible on an ultrasound scan
4. An undisturbed ectopic pregnancy and a serum human chorionic gonadotropins level of 5,000 IU/litre or more
5. intrauterine pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
determine efficacy of the aromatase inhibitor and Gnrh antagonist to achievement of resolution of ectopic pregnancy determined by serum hCG levels below laboratory immunoassay detection <15 IU/l.Results will be statistically analyzed,then evaluated . | 3 months

IPD SHARING:
Plan to Share IPD: Yes